CLINICAL TRIAL: NCT02076009
Title: Phase 3 Study Comparing Daratumumab, Lenalidomide, and Dexamethasone (DRd) vs Lenalidomide and Dexamethasone (Rd) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Comparing Daratumumab, Lenalidomide, and Dexamethasone With Lenalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103663; 54767414MMY3003 (Other: Janssen Research & Development, LLC); 2013-005525-23 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Daratumumab; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daratumumab + lenalidomide + dexamethasone (Experimental): During each 28-day treatment cycle, participants will receive daratumumab, lenalidomide, and dexamethasone.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Lenalidomide + dexamethasone (Active Comparator): During each 28-day treatment cycle, participants will receive lenalidomide and dexamethasone.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 16mg/kg will be administered as an intravenous (IV) infusion (into the vein) as per the following schedule: once a week during treatment cycles 1 and 2; every 2 weeks during treatment cycles 3 to 6; and every 4 weeks for cycles 7 and onwards. Following amendment 8, participants receiving daratumumab IV have the option to switch to daratumumab subcutaneous (SC) 1800 mg/dose until documented progression, unacceptable toxicity, or the end of study on Day 1 of any cycle, at the discretion of the investigator.
  Arms: Daratumumab + lenalidomide + dexamethasone
Drug: Lenalidomide — Lenalidomide will be administered at a dose of 25 mg orally (by mouth) on Days 1 through 21 of each treatment cycle.
Drug: Dexamethasone — Dexamethasone (or equivalent in accordance with local standards) will be administered as a total dose of 40 mg weekly (or 20 mg weekly for participants > 75 years old or with a body mass index < 18.5).

SUMMARY:
The purpose of this study is to compare the effectiveness of daratumumab when combined with lenalidomide and dexamethasone (DRd) to that of lenalidomide and dexamethasone (Rd), in terms of progression-free survival in participants with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a randomized (participants will be assigned by chance to study treatments), open-label (all participants and study personnel will know the identity of the study treatments), active-controlled (none of the study treatments are placebo), parallel-group (both treatment arms will run at the same time), multicenter study. In this study, daratumumab, lenalidomide, and low-dose dexamethasone (DRd) will be compared with lenalidomide and low dose dexamethasone (Rd) in participants with relapsed or refractory multiple myeloma. Participants will be randomized in a 1:1 ratio to receive either DRd or Rd. The study will include a Screening Phase, a Treatment Phase (involving treatment cycles of approximately 28 days in length), and a Follow-up Phase. The Treatment Phase will extend from the administration of the first dose of study medication until disease progression or unacceptable toxicity. Participants will also discontinue study treatment if: they become pregnant; have their dose held for more than 28 days (or if 3 consecutive planned doses of daratumumab are missed for reasons other than toxicity); or for safety reasons (for example, adverse event). The Follow-up Phase will begin at the end of treatment and will continue until death, loss to follow-up, consent withdrawal for study participation, or the final overall survival (OS) analysis, whichever occurs first. Eligible participants from Rd group who have had sponsor confirmed disease progression will be offered the option for treatment with daratumumab monotherapy (of 28 days cycle). The primary endpoint will be progression-free survival (PFS). Analysis of the primary endpoint was performed at a pre-specified point determined by PFS events with a clinical cutoff of March 7, 2016 when 169 events of death or progression had occurred. The end of study is anticipated at approximately 6 years after the last participant is randomized. Blood and urine samples will be obtained at time points during the study, together with bone marrow aspirates/biopsies and skeletal surveys. Participant safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented multiple myeloma and measurable disease
* Must have received at least 1 prior line of therapy for multiple myeloma and achieved a response (partial response or better) to at least one prior regimen
* Must have documented evidence of progressive disease as defined by the International Myeloma Working Group criteria on or after their last regimen
* Must have an Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2
* If a participant has received subsequent anticancer therapy (salvage therapy), the participant must have a "wash-out period" defined as 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the planned start date of daratumumab monotherapy. The only exception is the emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 milligram per day for a maximum of 4 days) before Daratumumab monotherapy

Exclusion Criteria:

* Has received any of the following therapies: daratumumab or other anti-CD38 therapies
* Has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment
* Disease shows evidence of refractoriness or intolerance to lenalidomide or if previously treated with a lenalidomide-containing regimen the participant is excluded if he or she discontinued due to any adverse event related to prior lenalidomide treatment
* Has received autologous stem cell transplantation within 12 weeks before the date of randomization, or previously received an allogenic stem cell transplant (regardless of timing), or planning to undergo a stem cell transplant prior to progression of disease
* History of malignancy (other than multiple myeloma) within 5 years before the first dose of daratumumab monotherapy (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or breast, or other non-invasive lesion, that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (145):
- United States (23):
  - Little Rock, Arkansas
  - Gainesville, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Bethesda, Maryland
  - Columbia, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Eugene, Oregon
  - Spartanburg, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Fairfax, Virginia
- Australia (6):
  - Camperdown
  - Geelong
  - Heidelberg
  - Malvern
  - South Brisbane
  - Southport
- Belgium (7):
  - Anderlecht
  - Antwerp
  - Edegem
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Denmark (3):
  - Copenhagen
  - Odense
  - Vejle
- France (12):
  - Argenteuil
  - Caen
  - Lille
  - Limoges
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rennes
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Berlin
  - Bonn
  - Cologne
  - Hamburg
  - Hamm
  - Heidelberg
  - Jena
  - Karlsruhe
  - Koblenz
  - Saarbrücken
  - Villingen-Schwenningen
- Athens Attica, Greece
- Israel (7):
  - Haifa
  - Jerusalem
  - Nahariya
  - Netanya
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Japan (15):
  - Hitachi
  - Kanazawa
  - Kobe
  - Kurume
  - Matsuyama
  - Nagoya
  - Narita
  - Ohgaki
  - Okayama
  - Osaka
  - Sendai
  - Shibukawa
  - Shibuya City
  - Tachikawa
  - Tokyo
- Netherlands (4):
  - Amsterdam
  - Rotterdam
  - Utrecht
  - Zwolle
- Poland (8):
  - Brzozów
  - Chorzów
  - Gdansk
  - Legnica
  - Lublin
  - Poznan
  - Słupsk
  - Wroclawa
- Russia (9):
  - Dzerzhinsk
  - Moscow
  - Nizhny Novgorod
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Syktyvkar
  - Yekaterinburg
- South Korea (3):
  - Gyeonggi-do
  - Incheon
  - Seoul
- Spain (7):
  - Badalona
  - Barcelona
  - La Laguna (Santa Cruz de Tenerife)
  - Madrid
  - Pamplona
  - Salamanca
  - Seville
- Sweden (7):
  - Falun
  - Gothenburg
  - Helsingborg
  - Huddinge
  - Lund
  - Stockholm
  - Uppsala
- Taiwan (5):
  - Changhua
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (7):
  - Birmingham
  - Leeds
  - London
  - Oxford
  - Southampton
  - Surrey
  - Wolverhampton

REFERENCES:
- [Derived] Almansour SA, Alqudah MAY, Abuhelwa Z, Al-Shamsi HO, Alhuraiji A, Semreen MH, Bustanji Y, Alzoubi KH, Modi ND, Mckinnon RA, Sorich MJ, Hopkins AM, Abuhelwa AY. Antithrombotic utilization, adverse events, and associations with treatment outcomes in multiple myeloma: pooled analysis of three clinical trials. Ther Adv Med Oncol. 2024 Sep 2;16:17588359241275387. doi: 10.1177/17588359241275387. eCollection 2024. PMID 39229471
- [Derived] Spencer A, Moreau P, Mateos MV, Goldschmidt H, Suzuki K, Levin MD, Sonneveld P, Orlowski RZ, Yoon SS, Usmani SZ, Weisel K, Reece D, Ahmadi T, Pei H, Mayo WG, Gai X, Carey J, Bartlett JB, Carson R, Dimopoulos MA. Daratumumab for patients with myeloma with early or late relapse after initial therapy: subgroup analysis of CASTOR and POLLUX. Blood Adv. 2024 Jan 23;8(2):388-398. doi: 10.1182/bloodadvances.2023010579. PMID 38048391
- [Derived] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Ahmadi T, Qin X, Garvin Mayo W, Gai X, Carey J, Carson R, Moreau P. Overall Survival With Daratumumab, Lenalidomide, and Dexamethasone in Previously Treated Multiple Myeloma (POLLUX): A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2023 Mar 10;41(8):1590-1599. doi: 10.1200/JCO.22.00940. Epub 2023 Jan 4. PMID 36599114
- [Derived] Cavo M, San-Miguel J, Usmani SZ, Weisel K, Dimopoulos MA, Avet-Loiseau H, Paiva B, Bahlis NJ, Plesner T, Hungria V, Moreau P, Mateos MV, Perrot A, Iida S, Facon T, Kumar S, van de Donk NWCJ, Sonneveld P, Spencer A, Krevvata M, Heuck C, Wang J, Ukropec J, Kobos R, Sun S, Qi M, Munshi N. Prognostic value of minimal residual disease negativity in myeloma: combined analysis of POLLUX, CASTOR, ALCYONE, and MAIA. Blood. 2022 Feb 10;139(6):835-844. doi: 10.1182/blood.2021011101. PMID 34289038
- [Derived] Plesner T, Dimopoulos MA, Oriol A, San-Miguel J, Bahlis NJ, Rabin N, Suzuki K, Yoon SS, Ben-Yehuda D, Cook G, Goldschmidt H, Grosicki S, Qin X, Fastenau J, Garvin W, Carson R, Renaud T, Gries KS. Health-related quality of life in patients with relapsed or refractory multiple myeloma: treatment with daratumumab, lenalidomide, and dexamethasone in the phase 3 POLLUX trial. Br J Haematol. 2021 Jul;194(1):132-139. doi: 10.1111/bjh.17435. Epub 2021 Apr 6. PMID 33822368
- [Derived] Avet-Loiseau H, San-Miguel J, Casneuf T, Iida S, Lonial S, Usmani SZ, Spencer A, Moreau P, Plesner T, Weisel K, Ukropec J, Chiu C, Trivedi S, Amin H, Krevvata M, Ramaswami P, Qin X, Qi M, Sun S, Qi M, Kobos R, Bahlis NJ. Evaluation of Sustained Minimal Residual Disease Negativity With Daratumumab-Combination Regimens in Relapsed and/or Refractory Multiple Myeloma: Analysis of POLLUX and CASTOR. J Clin Oncol. 2021 Apr 1;39(10):1139-1149. doi: 10.1200/JCO.20.01814. Epub 2021 Jan 29. PMID 33513030
- [Derived] Mateos MV, Spencer A, Nooka AK, Pour L, Weisel K, Cavo M, Laubach JP, Cook G, Iida S, Benboubker L, Usmani SZ, Yoon SS, Bahlis NJ, Chiu C, Ukropec J, Schecter JM, Qin X, O'Rourke L, Dimopoulos MA. Daratumumab-based regimens are highly effective and well tolerated in relapsed or refractory multiple myeloma regardless of patient age: subgroup analysis of the phase 3 CASTOR and POLLUX studies. Haematologica. 2020 Jan 31;105(2):468-477. doi: 10.3324/haematol.2019.217448. Print 2020. PMID 31221782
- [Derived] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Komarnicki M, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Lisby S, Khokhar NZ, O'Rourke L, Chiu C, Qin X, Guckert M, Ahmadi T, Moreau P; POLLUX Investigators. Daratumumab, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Oct 6;375(14):1319-1331. doi: 10.1056/NEJMoa1607751. PMID 27705267

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide, Low-dose Dexamethasone (Rd): Participants received lenalidomide at a dose of 25 milligrams (mg) orally on Day 1 through Day 21 of each 28-day treatment cycle and low-dose dexamethasone at a total dose of 40 mg weekly (or 20 mg weekly for participants greater than [>] 75 years old or with a body mass index less than [<] 18.5 kilograms per meter square [kg/m^2]).
- Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd): Participants received daratumumab 16 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion once a week during treatment cycles 1 and 2 (for 8 weeks, each 28-day cycle); every 2 weeks during treatment cycles 3 to 6 (for 16 weeks, each 28-day cycle); once only on Day 1 during treatment cycles 7 onwards (for every 4 weeks). Lenalidomide was administered at a dose of 25 mg orally on Day 1 through Day 21 of each 28-day treatment cycle and low-dose dexamethasone was administered at a total dose of 40 mg weekly (or 20 mg weekly for participants >75 years old or with a body mass index < 18.5 kg/m^2).
Period: Overall Study
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Started | 283 | 286
Treated (Safety Population) | 281 | 283
Completed | 0 | 0
Not Completed | 283 | 286
Not completed — Death | 172 | 153
Not completed — Withdrawal by Subject | 16 | 12
Not completed — Lost to Follow-up | 4 | 2
Not completed — Progressive Disease | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — End of data collection | 90 | 118

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd) | Total
Number analyzed (Participants) | 283 | 286 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.84) | 64.4 (9.03) | 64.4 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 113 | 232
  Male | 164 | 173 | 337
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 9 | 9 | 18
  Belgium | 10 | 12 | 22
  Canada | 17 | 17 | 34
  Denmark | 7 | 10 | 17
  France | 36 | 21 | 57
  Germany | 7 | 11 | 18
  Greece | 8 | 11 | 19
  Israel | 20 | 19 | 39
  Japan | 15 | 21 | 36
  Korea, Republic of | 20 | 20 | 40
  Netherlands | 3 | 1 | 4
  Poland | 13 | 15 | 28
  Russian Federation | 30 | 18 | 48
  Spain | 25 | 26 | 51
  Sweden | 15 | 16 | 31
  Taiwan, Province of China | 9 | 11 | 20
  United Kingdom | 24 | 27 | 51
  United States | 15 | 21 | 36
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of following 3 stages - Stage I: serum beta2-microglobulin less than (<) 3.5 milligram per liter (mg/L) and albumin greater than or equal to (>=) 3.5 gram per 100 milliliter (g/100 ml); Stage II: neither stage I nor stage III and Stage III: serum beta2-microglobulin >= 5.5 mg/L.
  Participants
    I | 140 | 137 | 277
    II | 86 | 93 | 179
    III | 57 | 56 | 113
No. of Prior Lines of Therapy [Count of Participants; unit: Participants]
  1 | 146 | 149 | 295
  2 | 80 | 85 | 165
  3 | 38 | 38 | 76
  >3 | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS: duration from date of randomization to either progressive disease (PD)/death, whichever occurred first. PD: defined as meeting any 1 of following criteria: Increase of greater than equal to (>=)25 percent(%) in level of serum M-protein from lowest response value and absolute increase must be >=0.5 gram per deciliter (g/dL); Increase of >=25% in 24-hours(h) urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24h; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved free light chain (FLC) levels from lowest response value and absolute increase must be >10 mg/dL; Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) attributed solely to plasma cell (PC) proliferative disorder.
Time Frame: From randomization to either disease progression or death whichever occurs first (up to 21 months)
Population: Intent-to-treat (ITT) analysis set included all participants who were randomly assigned to the daratumumab, lenalidomide, dexamethasone (DRd) or lenalidomide, low-dose dexamethasone (Rd) group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 283 | 286
months | 18.43 [13.86 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to short follow-up by participants. | NA [NA to NA] — Median and 95% CI was not estimable due to short follow-up by participants.

2. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined as time from date of randomization to date of first documented evidence of progressive disease (PD). PD was defined as meeting any one of following criteria: Increase of >=25% in level of serum M-protein from lowest response value and absolute increase must be >=0.5 g/dL; Increase of >=25% in 24-hour urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24hours; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved free light chain (FLC) levels from lowest response value and absolute increase must be >10 milligram per deciliter (mg/dL); Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to plasma cell (PC) proliferative disorder.
Time Frame: From randomization to disease progression (up to 21 months)
Population: ITT analysis set included all participants who were randomly assigned to the DRd or Rd group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 283 | 286
months | 18.43 [14.78 to NA] — Upper limit of 95% CI was not estimable due to short follow-up. | NA [NA to NA] — Median and 95% CI was not estimable due to short follow-up.

3. Secondary Outcome: Percentage of Participants Who Achieved Very Good Partial Response (VGPR) or Better
Description: VGPR or better is defined as the percentage of participants who achieved VGPR, complete response (CR) and stringent complete response (sCR) according to the International Myeloma Working Group criteria (IMWG). IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >90% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required; CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4 color flow cytometry.
Time Frame: From randomization to disease progression (up to 21 months)
Population: Response-evaluable set included participants who have a confirmed diagnosis of multiple myeloma and measurable disease and must have received at least 1 administration of study treatment and have at least 1 post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 276 | 281
percentage of participants | 44.2 [38.3 to 50.3] | 75.8 [70.4 to 80.7]

4. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: Minimal residual disease was assessed for all participants who achieved a complete response (CR) or stringent complete response (sCR). CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4 color flow cytometry. The MRD negativity rate was defined as the percentage of participants who had negative MRD assessment at any time point after the first dose of study drugs by evaluation of bone marrow aspirates or whole blood at 10^ minus (-) 4, 10^-5, 10^-6 threshold.
Time Frame: From randomization to the date of first documented evidence of PD (up to 87.5 months)
Population: ITT analysis set included all participants who were randomly assigned to the DRd or Rd group.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 283 | 286
percentage of participants
  MRD negative rate (10^-4) | 10.2 [7.0 to 14.4] | 40.6 [34.8 to 46.5]
  MRD negative rate (10^-5) | 6.7 [4.1 to 10.3] | 33.2 [27.8 to 39.0]
  MRD negative rate (10^-6) | 1.8 [0.6 to 4.1] | 13.3 [9.6 to 17.8]

5. Secondary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants who achieved a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria, during or after study treatment. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From randomization to disease progression (up to 21 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 276 | 281
percentage of participants | 76.4 | 92.9

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the date of randomization to the date of the participant's death.
Time Frame: From randomization to date of death due to any cause (up to 87.5 months)
Population: ITT analysis set included all participants who were randomly assigned to the DRd or Rd group. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 175 | 153
months | 51.84 [43.99 to 60.02] | 67.58 [53.13 to 80.53]

7. Secondary Outcome: Time to Response
Description: Time to response was defined as the time between the date of randomization and the first efficacy evaluation that the participant met all criteria for partial response (PR) or better.
Time Frame: From randomization up to first documented CR or PR (up to 21 months)
Population: Response-evaluable set is defined as participants who have a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit. In addition, participants must have received at least 1 administration of study treatment and have at least 1 post baseline disease assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 276 | 281
months | 1.3 [1.1 to 1.9] | 1.0 [1.0 to 1.1]

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for participants with confirmed response (PR or better) as time between first documentation of response and disease progression/death due to PD, whichever occurs first. PD was defined as meeting any one of following criteria: Increase of >=25% in level of serum M-protein from lowest response value and absolute increase must be >=0.5g/dL; Increase of >=25% in 24-hour urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200mg/24hours; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved FLC levels from lowest response value and absolute increase must be >10mg/dL; Definite increase in size of existing bone lesions/soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From randomization to the date of first documented evidence of PD (up to 21 months)
Population: Response-evaluable set included participants who have a confirmed diagnosis of multiple myeloma and measurable disease and must have received at least 1 administration of study treatment and have at least 1 post baseline disease assessment. Here 'N' signifies number of participants who had PR or better response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 211 | 261
months | 17.4 [17.4 to NA] — Upper limit of 95% CI was not estimable due to high censoring rate and lesser number of responders who progressed. | NA [NA to NA] — Median and 95% CI was not estimable due to high censoring rate and lesser number of responders who progressed.

9. Secondary Outcome: Time to Subsequent Anticancer Treatment
Description: Time to subsequent anticancer treatment was defined as the time from randomization to the start of subsequent anticancer treatment or death due to progressive disease (PD), whichever occurs first.
Time Frame: From randomization to date of start of subsequent anticancer treatment or death due to PD, whichever occured first (up to 87.5 months)
Population: ITT analysis set included all participants who were randomly assigned to the DRd or Rd group, and who started subsequent anticancer therapy or died due to progressive disease, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Number analyzed (Participants) | 212 | 138
months | 23.1 [18.6 to 26.3] | 69.3 [49.7 to 82.8]

ADVERSE EVENTS:
Time Frame: From randomization up to 30 days after last dose of study treatment (up to 87.5 months)
Description: Safety analysis set included all randomized participants who had at least 1 administration of any study treatment (partial or complete).
Arm/Group | Lenalidomide, Low-dose Dexamethasone (Rd) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd)
Serious Adverse Events (participants affected / at risk) | 148/281 | 205/283
Other Adverse Events (participants affected / at risk) | 268/281 | 278/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Low-dose Dexamethasone (Rd) (N=281) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd) (N=283)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 13
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 5
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 3
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Pericarditis (Cardiac disorders) | 1 | 2
Right ventricular failure (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 4
Keratitis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 2
Visual field defect (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 8
Diverticular perforation (Gastrointestinal disorders) | 0 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Generalised oedema (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 3 | 3
Pain (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 13
Sudden death (General disorders) | 1 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Arthritis bacterial (Infections and infestations) | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 10
Bronchitis bacterial (Infections and infestations) | 0 | 1
Brucellosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 3
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 4
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 3
Gastrointestinal infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 6 | 3
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Infective spondylitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 7 | 12
Intervertebral discitis (Infections and infestations) | 0 | 1
Keratitis fungal (Infections and infestations) | 1 | 0
Legionella infection (Infections and infestations) | 0 | 1
Listeria sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 14
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 3
Nocardiosis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 0
Otitis externa (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 1
Parotitis (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 32 | 48
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia haemophilus (Infections and infestations) | 0 | 2
Pneumonia influenzal (Infections and infestations) | 0 | 7
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 3
Respiratory tract infection (Infections and infestations) | 2 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 8 | 7
Septic shock (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 7
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 3
Uterine abscess (Infections and infestations) | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Posterior capsule rupture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
Diagnostic procedure (Investigations) | 1 | 0
Influenza B virus test positive (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 2 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 5
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 1
Depressive symptom (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 11 | 8
Azotaemia (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 5 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Loss of personal independence in daily activities (Social circumstances) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Embolism (Vascular disorders) | 0 | 1
Femoral artery embolism (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Low-dose Dexamethasone (Rd) (N=281) | Daratumumab, Lenalidomide, Low-dose Dexamethasone (DRd) (N=283)
Anaemia (Blood and lymphatic system disorders) | 117 | 118
Leukopenia (Blood and lymphatic system disorders) | 23 | 29
Lymphopenia (Blood and lymphatic system disorders) | 17 | 20
Neutropenia (Blood and lymphatic system disorders) | 136 | 185
Thrombocytopenia (Blood and lymphatic system disorders) | 90 | 92
Atrial fibrillation (Cardiac disorders) | 9 | 17
Tachycardia (Cardiac disorders) | 2 | 16
Cataract (Eye disorders) | 35 | 59
Vision blurred (Eye disorders) | 17 | 28
Abdominal pain (Gastrointestinal disorders) | 16 | 30
Abdominal pain upper (Gastrointestinal disorders) | 13 | 29
Constipation (Gastrointestinal disorders) | 77 | 94
Diarrhoea (Gastrointestinal disorders) | 105 | 169
Dyspepsia (Gastrointestinal disorders) | 9 | 29
Nausea (Gastrointestinal disorders) | 53 | 86
Stomatitis (Gastrointestinal disorders) | 6 | 19
Toothache (Gastrointestinal disorders) | 10 | 17
Vomiting (Gastrointestinal disorders) | 19 | 65
Asthenia (General disorders) | 47 | 59
Chills (General disorders) | 9 | 22
Fatigue (General disorders) | 87 | 119
Influenza like illness (General disorders) | 20 | 27
Non-cardiac chest pain (General disorders) | 5 | 18
Oedema peripheral (General disorders) | 50 | 72
Pyrexia (General disorders) | 40 | 71
Bronchitis (Infections and infestations) | 45 | 60
Conjunctivitis (Infections and infestations) | 6 | 19
Gastroenteritis (Infections and infestations) | 9 | 25
Influenza (Infections and infestations) | 17 | 34
Lower respiratory tract infection (Infections and infestations) | 12 | 22
Nasopharyngitis (Infections and infestations) | 62 | 100
Pneumonia (Infections and infestations) | 27 | 51
Respiratory tract infection (Infections and infestations) | 29 | 38
Rhinitis (Infections and infestations) | 5 | 23
Sinusitis (Infections and infestations) | 13 | 27
Upper respiratory tract infection (Infections and infestations) | 74 | 123
Urinary tract infection (Infections and infestations) | 26 | 30
Contusion (Injury, poisoning and procedural complications) | 12 | 25
Fall (Injury, poisoning and procedural complications) | 12 | 24
Alanine aminotransferase increased (Investigations) | 14 | 19
Blood creatinine increased (Investigations) | 17 | 16
Weight decreased (Investigations) | 13 | 31
Decreased appetite (Metabolism and nutrition disorders) | 36 | 50
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 34
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 58
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 75
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 76
Bone pain (Musculoskeletal and connective tissue disorders) | 16 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 61 | 87
Muscular weakness (Musculoskeletal and connective tissue disorders) | 26 | 29
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 24 | 32
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 22
Neck pain (Musculoskeletal and connective tissue disorders) | 13 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 47
Dizziness (Nervous system disorders) | 30 | 35
Headache (Nervous system disorders) | 23 | 56
Hypoaesthesia (Nervous system disorders) | 9 | 18
Neuropathy peripheral (Nervous system disorders) | 18 | 25
Paraesthesia (Nervous system disorders) | 12 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 40
Tremor (Nervous system disorders) | 26 | 28
Anxiety (Psychiatric disorders) | 13 | 25
Depression (Psychiatric disorders) | 9 | 29
Insomnia (Psychiatric disorders) | 65 | 80
Renal impairment (Renal and urinary disorders) | 15 | 33
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 65
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 23
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 26
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 21
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 18
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 34
Rash (Skin and subcutaneous tissue disorders) | 36 | 51
Haematoma (Vascular disorders) | 6 | 15
Hypertension (Vascular disorders) | 22 | 31
Hypotension (Vascular disorders) | 9 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.